CLINICAL TRIAL: NCT05045235
Title: Optimization of Drug Prescriptions in the Care Pathway for the Elderly, With the Final Objective of Reducing the Iatrogenic Risk.
Acronym: IATROPREV
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0158
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Iatrogenic Effect; Prescription; Follow-up; Consultation
Keywords: iatrogenic; prescription; follow-up; consultation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The IATROPREV project is an organizational innovation experimentation project, carried out in Hauts-de-France by the University hospitals of Amiens and Lille, the ARS and the URPS Doctors and Pharmacists of Hauts-de-France and following to the social security financing law of 2018, allowing experimentation with new organizations in the health sector, according to article 51. The objectives of this course are to improve the relevance of prescription in elderly people with multiple drugs as well as, the coordination of care between the city and the hospital through the sharing of information and the establishment of multi-professional consultations between the various care actors.

ELIGIBILITY:
Inclusion Criteria:

* patient hospitalized in the geriatric medicine department
* Potential involvement of a drug in hospitalization or potential or proven iatrogenic event during hospitalization;
* Numerous therapeutic modifications (3 or more);
* Drug interaction or introction of a new drug with one or more drug interactions;
* Medicinal product with a narrow therapeutic marge drug requiring close monitoring.

Exclusion Criteria:

* patient non hospitalized in the geriatric medicine department

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient hospitalized in the geriatric medicine department with olymedicated drugs
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change of side effect number in ederly with polymedicated drugs | up to 4 years
  Change of side effect number in ederly with polymedicated drugs

CONTACTS AND LOCATIONS:
Locations (1):
- Amiens University Hospital, Amiens, France

IPD SHARING:
Plan to Share IPD: No